CLINICAL TRIAL: NCT01156129
Title: Interventions to Decrease the Impact of Post-Operative Ileus After Liver Transplant or Resection Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0228-10-FB
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Ileus
Keywords: liver transplant; liver resection
MeSH Terms: conditions — Ileus | interventions — Dioctyl Sulfosuccinic Acid; Magnesium Hydroxide; Bisacodyl; Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: Standard therapy (use of medications) (Active Comparator): stool softener
  Interventions: Drug: stool softener
- Arm B: Acupressure bracelets (Experimental): device - Biobands
  Interventions: Device: Arm B: Acupressure bracelet
- Arm C (Experimental): Sugar free gum
  Interventions: Dietary Supplement: sugar free gum

INTERVENTIONS:
Drug: stool softener — ducosate sodium, Milk of Magnesia, dulcolax
  Other Names: Milk of Magnesia, Dulcolax
  Arms: Arm A: Standard therapy (use of medications)
Device: Arm B: Acupressure bracelet — Bioband
  Other Names: Bioband
  Arms: Arm B: Acupressure bracelets
Dietary Supplement: sugar free gum — Orbit
  Other Names: generic
  Arms: Arm C

SUMMARY:
This is a randomized controlled trial to assess ways to address post-operative ileus (POI) in adult patients on the liver transplant service undergoing either liver transplant or resection surgery. Patient who speak and understand English will be randomized into one of three groups including a.)control group receiving standard therapy for post-operative ileus, b.)group receiving standard therapy and acupressure bracelets, and c.)group receiving standard therapy and sugar free gum four times daily.

DETAILED DESCRIPTION:
Any patient undergoing liver transplant or resection surgery will be asked to participate in the study and assigned to a control or investigational group. Pertinent information will be collected from the medical record including gender, age in years, diagnosis, type of surgery, length of stay, medications used for pain or nausea, and first bowel movement. The subjects will also be asked to keep a journal of their bowel habits, signs and symptoms of gastrointestinal distress/post-operative ileus, use of medications, first bowel movement, satisfaction with bowel management and any additional comments.

Aims of the study are to determine the effectiveness of the three arms of this trial for the resolution of POI as noted by first post-operative bowel movement; to determine if there is a difference in the length of stay based on the interventions; and to determine if there is a difference in patient satisfaction based on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 years or older who speak and read English and have had a liver transplant or liver resection surgery

Exclusion Criteria:

* Patients less than 19 years of age having liver transplant or liver resection surgery
* Non-English speaking
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
Timing of first post operative bowel movement | Days post operative
  First bowel movement

SECONDARY OUTCOMES:
Length of hospital stay | Time from admission to discharge post surgery
  Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Laurel W Williams, MSN,RN, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States